CLINICAL TRIAL: NCT02018796
Title: Acceptability and Feasibility of a Simplified Medical Abortion Regimen in Kazakhstan: A Study of 600 µg Sublingual Misoprostol Following 200 mg Mifepristone for Abortion up to 70 Days Gestation
Brief Title: Mifepristone and Misoprostol for the Termination of Pregnancy up to 70 Days' Gestation in Kazakhstan
Status: Completed | Type: Observational
Sponsor: Gynuity Health Projects (Other)
Responsible Party: Sponsor
Other Study IDs: 1011
Record Dates: First submitted 2013-12-10; First posted 2013-12-23 (Estimated); Last update posted 2015-08-13 (Estimated); Status verified 2015-08

CONDITIONS: Complete Abortion
MeSH Terms: interventions — Mifepristone; Misoprostol

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Women seeking medical abortion: Women with pregnancies less than 71 days gestation seeking medical abortion. Women who choose to participate in the study will be administered 200 mifepristone, followed 24 to 48 hours later by 600 mcg misoprostol.
  Interventions: Drug: Mifepristone, misoprostol

INTERVENTIONS:
Drug: Mifepristone, misoprostol — 200 mifepristone, followed 24 to 48 hours later by 600 mcg misoprostol

SUMMARY:
The study will be conducted in 4 sites and will examine how a simplified outpatient medical abortion procedure using mifepristone and misoprostol, with the option to take mifepristone at a place of woman's choosing, works in Kazakhstan. The investigators intend to demonstrate the efficacy of oral administration of 200 mg mifepristone and sublingual administration of 600 µg misoprostol with gestations through 70 days, as well as the acceptability of this method. Research questions include:

1. What is the efficacy of regimen of 200 mg mifepristone, followed 24 to 48 hours later by 600 µg sublingual misoprostol and used in gestations of up to 70 days?
2. Is medical abortion procedure consisting of two visits acceptable to women in Kazakhstan?
3. Are the side effects associated with sublingual use of misoprostol acceptable to women?
4. When given a choice, do women prefer to take mifepristone in the clinic or at a place of their choosing?

ELIGIBILITY:
Inclusion Criteria:

* Have an intrauterine pregnancy consistent with gestational age less than 71 days;
* Be able to understand and willing to sign a consent form;
* Be eligible for medical abortion according to the clinician's assessment;
* Be able to return to the clinic and able to contact study staff or emergency medical services, if needed;
* Be willing to provide an address and/or telephone number for purposes of follow-up;
* Agree to comply with the study procedures and visit schedule.

Exclusion Criteria:

* Confirmed or suspected ectopic pregnancy or undiagnosed adnexal mass;
* Chronic renal failure;
* Concurrent long-term corticosteroid therapy;
* History of allergy to mifepristone, or misoprostol or another prostaglandin;
* History of hemorrhagic disorders or concurrent anticoagulant therapy;
* History of inherited porphyrias;
* Intrauterine device in place (must be removed before mifepristone is administered).

Sex: Female | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: Women seeking an abortion at participating study sites
Sampling Method: Non-Probability Sample
Enrollment: 290 (Actual)
Dates: Start 2013-10; Primary Completion 2014-12 (Actual); Study Completion 2014-12 (Actual)

PRIMARY OUTCOMES:
Rate of successful abortion | 2 weeks after mifepristone administration

SECONDARY OUTCOMES:
Satisfaction with method | 2 weeks or up to 30 days after mifepristone administration

OTHER OUTCOMES:
Number of days missed work/school for women choosing mifepristone administration outside the clinic and those who choose its administration at the clinic | 2 weeks after mifepristone administration
Side effects | 2 weeks after mifepristone administration
Acceptability of the side effects and of sublingual administration | 2 weeks after mifepristone administration
Complications, including heavy bleeding or infection requiring additional treatment | 2 weeks after mifepristone administration

CONTACTS AND LOCATIONS:
Overall Officials: Beverly Winikoff, MD, PhD, Principal Investigator — Gynuity Health Projects; Mariya Bashkirova, MD, Principal Investigator — Almaty City Policlinic No 19, Almaty, Kazakhstan; Tina Kan, MD, Principal Investigator — Almaty City Policlinic No. 9, Almaty, Kazakhstan; Gulnar Mukazhanova, MD, Principal Investigator — Consultation and Diagnostics Department, Regional Perinatal Center, Astana, Kazakhstan; Oksana Kolyadinova, MD, Principal Investigator — Consultation and Diagnostics Department, City Maternity House, Astana, Kazakhstan; Galina Grebennikova, MD, Study Director — Kazakhstan Association on Sexual and Reproductive Health; Tamar Tsereteli, MD, MSc, PhD, Study Director — Gynuity Health Projects
Locations (4):
- Kazakhstan (4):
  - Almaty City Policlinic No. 19, Almaty
  - Almaty City Policlinic No. 9, Almaty
  - Consultation and Diagnostics Department of the City Maternity House, Astana
  - Consultation and Diagnostics Department of the Regional Perinatal Center No. 2, Astana

REFERENCES:
- [Derived] Platais I, Tsereteli T, Grebennikova G, Lotarevich T, Winikoff B. Prospective study of home use of mifepristone and misoprostol for medical abortion up to 10weeks of pregnancy in Kazakhstan. Int J Gynaecol Obstet. 2016 Sep;134(3):268-71. doi: 10.1016/j.ijgo.2016.02.018. Epub 2016 May 26. PMID 27352735
- See also: Kazakhstan Association on Sexual and Reproductive Health — http://www.kmpakaz.org/